CLINICAL TRIAL: NCT00301054
Title: Preventing Anemia in Children (6months-30months) in a Malaria Endemic Rural Area in Ghana - A Randomized Double Blind Study
Brief Title: Study on Preventing Anemia in Children in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ghana Health Services (Other Government)
Collaborators: Netherlands Overseas Agency (Ambiguous)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2003/GD/23
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2005-07

CONDITIONS: Anaemia in Children
Keywords: Anaemia; Malaria; Rural Area in Ghana
MeSH Terms: conditions — Anemia; Malaria | interventions — ferrous sulfate; fanasil, pyrimethamine drug combination

INTERVENTIONS:
Drug: Ferrous sulphate
Drug: Sulphadoxine-Pyrimethamine

SUMMARY:
A study that seeks to establish an effective way of preventing anaemia in children at the community level using two known interventions - Iron supplementation and or antimalarial. Children recruited into the study will be assigned to four groups. Those receiving Placebo and Iron, those receiving Placebo and Antimalarial, those receiving Placebo and Antimalarial and those receiving double placebo. The children will be followed up over a period of nine months and their haemoglobin concentration, malaria parasites in their blood and their weight and height will be assessed.

DETAILED DESCRIPTION:
I. INTRODUCTION

Anaemia in children is a major problem in developing countries 1. Iron deficiency is believed to be the most common form of anaemia in children. In some countries fortification of some common foods for children with iron has led to a decrease in morbidity and mortality associated with iron deficiency anemia.2 In malaria endemic areas, anaemia in children is made worse by incidence of malaria.

Brief Background of the District

Berekum District is one of the thirteen administrative districts in the Brong Ahafo Region of Ghana it has a total surface area of 1094.2 sq.km. The estimated population based on the 2000 census with a growth rate of 2.5% is approximately 102,914 for the year 2004.Male to female ratio in the district is 1:1.1. The inhabitants are mainly Brongs with other ethnic groups from all over the country. 55.3% of the population live in the rural area.

II. PROBLEM ANALYSIS

Anaemia is recognised as a worldwide public health problem. It is estimated by the World Health Organization that the prevalence of anaemia defined by haemoglobin less than 11.0g/dl is about 33%.5 In Berekum District the prevalence of anaemia in children defined as haemoglobin concentration less than 10.0g/dl was found to be 80% in a nutritional survey carried out in communities in the district in 1994.6 Anaemia is one of the major causes of mortality in children under five years in Ghana.

III. AIMS AND OBJECTIVES OF THE STUDY

The aim of this study is to establish an effective way of preventing anaemia in children at the community level.

The specific objectives of the study are:

1. To determine the impact of weekly iron supplementation on the prevention of anaemia, increase in haemoglobin, growth parameters, and susceptibility to malaria (during and after treatment) in children 6-30months.
2. To determine the impact of monthly sulphadoxine-pyrimethamine administration on the prevention of anaemia, increase in haemoglobin, growth parameters, and susceptibility to malaria (during and after treatment) in children 6-30months.
3. To determine which of the interventions is more effective in preventing anaemia and increasing haemoglobin concentration in children aged 6-30months compared to placebo.
4. To determine if there is a synergistic effect in giving both iron and sulphadoxine-pyrimethamine in preventing anaemia in children aged 6-30months.
5. To find out the percentage of children who have adverse reaction when given Sulphadoxine-pyrimethamine.
6. To determine if there is a difference in the incidence of clinical cases of vaccine preventable diseases among the intervention groups compared to the placebo.

STUDY TYPE

This is a Randomized double blind placebo-controlled study which will try to assess the effectiveness of three interventions in preventing anaemia in the community.

STUDY POPULATION

The universe population is all children 6months - 30months who reside in any of the communities in Berekum District. The target population are children who are 6months- 30months living in the Berekum District who attend well baby clinic.

The study population will be the children who are between the ages 6months- 30months attending well baby clinic at twenty immunization sites in the district. Those who will attend child welfare clinic on the day the research team visit will be chosen if they fall within the age range and their mothers agree to let them take part in the study.

SAMPLING

Using 2x2 factorial design, a sample size of 189 per each of the four groups will be required to measure a difference in haemoglobin concentration between the groups within 0.5g/dl of the true value (alpha = 0.05). With an estimated drop out rate of 15% a total sample size of approximately 872 or 218 per group will be used.

The placebo group represents the child welfare service that is currently available for children in the district, and in the rest of the country, so little ethical concerns are raised in recruiting children into the placebo group. They will also be of help in determining if there is difference in the occurrence of clinical cases of three vaccine preventable diseases(measles, acute flaccid paralysis and whooping cough) among children in any of the intervention groups compared to the placebo group, which can be used as a proxy indicator of possible adverse EPI vaccines and interventions interaction.

An assumption is being made that since the district is very homogenous and consists mainly of one tribe predominantly, children selected at the various sites do not differ markedly from each other in terms of diet and exposure to other factors that might lead to anaemia. Furthermore, there is 98% child welfare attendance coverage in the District. Therefore, children attending child welfare clinics are quite representative of the community. Children at the twenty immunization/child welfare clinic sites in the district will randomly be assigned into one of the four study groups, after obtaining consent from their parents for them to be enrolled in the study. A simple randomization scheme will be utilized. Given the trial size, balance in treatment/placebo group sizes is anticipated. A recruitment questionnaire will be completed for all children recruited into the study.

INTERVENTIONS

The interventions that will be used are:

1. Weekly iron supplementation Iron (II) Sulphate tablet at dose of 2mg/kg body weight and monthly placebo resembling sulphadoxine-pyrimethamine tablet.
2. Weekly placebo resembling Iron (II) Sulphate tablet and monthly treatment with sulphadoxine-pyrimethamine according to body weight (¼ tablet for those < 5kg, ½ tablet for those 5-10 kg and 1 tablet for those 10-15kg.
3. Weekly iron supplementation Iron (II) Sulphate tablet at dose of 2mg/kg body weight and monthly Sulphadoxine-pyrimethamine tablet
4. Weekly placebo resembling iron (II) sulphate tablet and monthly placebo resembling sulphadoxine-pyrimethamine tablet

Interventions will be pre-packed and labelled with drug code numbers by the manufacturers. Children will randomly be assigned to a pre-packed drug by community health nurses working in the community. Community health nurses will not be aware of which intervention each child is receiving. Code as to what each child is on will be held in a seal and kept by the drug manufacturers, till data is ready for analysis. To ensure compliance, every week community health nurses will visit the communities and give the drugs to the children under direct observation.

FOLLOW-UP

The intervention will be given to the children for a period of 6months.Children will be followed up for another 3months post-intervention. Community Health Nurses will visit children weekly to assess cutaneous reactions and check axillary temperature. At baseline, 2months, 4months, 6months and 9months blood samples will be taken to measure haemoglobin concentration in g/dl to assess anaemia. Haemoglobin concentration will be measured twice for each child on each occasion. Malaria will be determined by looking at thick and thin blood film, which will be stained and read using standard procedure to look for asexual forms of P falciparum4. Children seen in the community by the community health nurses with axillary temperature above 37.5 Celsius without any complications will be treated with Chloroquine according to their weight; those with complicated malaria will be admitted to the ward. The project will pay for this treatment. Haemoglobin electrophoresis for sickle cell will be done using cellulose acetate. The weight and length of the children will be taken at baseline, 2months, 4months, 6months and 9months by the four community health nurses working at immunization sites.

V. PLAN FOR DATA ANALYSIS

Data will be analyzed using Epi 2000.Difference in Haemoglobin change between the groups over the period will be determined using the Student t-test at 95% confidence interval. Proportion of those with weight to age and length to age ratio between -2SD and +2SD and those with Plasmodium falciparum in thick peripheral blood film will be calculated. These two proportions will be compared between the two interventions and the placebo at the various time periods using Chi-square analysis; it will be determined where there is significance difference between the proportions of the interventions at 95% confidence interval compared to each other and compared to the placebo group. Average febrile episodes will be compared between the interventions and the placebo using ANOVA to determine significance difference at 95% confidence interval.

VI. ETHICAL ISSUES

Proposal for study will be submitted to the National committee for ethics in Research. Interventions that will be used have a long history of use and most of the side-effects are already known and have been documented. Giving Iron supplementation to children is a public health intervention that has been done in a lot of settings to prevent anaemia and found to be safe. Use of sulphadoxine-pyrimethamine in treating malaria is also very extensive especially in the Southern parts of Africa. Children will be closely monitored, and mothers will be required to report any adverse reactions that they notice. Children who appear to react adversely to any of the interventions will be dropped from the study. . Mothers' access to routine health services for their children will not be affected by mother's refusal to participate in this study.

Verbal informed consent will be obtained from mothers of chosen children.

ELIGIBILITY:
Inclusion Criteria:

* All children living in Berekum District who are between 6months- 30months

Exclusion Criteria:

* All Children living in Berekum District between 6months- 30months who are G6PD Deficient

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 872
Dates: Start 2005-06; Study Completion 2006-04

PRIMARY OUTCOMES:
Haemoglobin concentration, Blood Film for malaria parasitaemia, weight/height ratio

SECONDARY OUTCOMES:
Incidence of vaccine preventable diseases like measles whooping cough(pertussis)

CONTACTS AND LOCATIONS:
Overall Officials: ANTHONY A OFOSU, MBChB, MPH, Principal Investigator — GHANA HEALTH SERVICE BEREKUM DISTRICT; DONNA M DENNO, MD, PAEDS, Study Director — UNIVERSITY OF WASHINGTON MEDICAL CENTER, SEATTLE, USA
Locations (1):
- District Health Directorate, Berekum, Brong- Ahafo, Ghana

REFERENCES:
- [Background] Alonzo Gonzalez M, Menendez C, Font F, Kahigwa E, Kimario J, Mshinda H, Tanner M, Bosch-Capblanch X, Alonso PL. Cost-effectiveness of iron supplementation and malaria chemoprophylaxis in the prevention of anaemia and malaria among Tanzanian infants. Bull World Health Organ. 2000;78(1):97-107. PMID 10686744
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597